CLINICAL TRIAL: NCT03289039
Title: A Phase 2 Study of Neratinib With or Without Fulvestrant in HER2-Positive, ER-Positive Metastatic Breast Cancer
Brief Title: Neratinib +/- Fulvestrant in HER2+, ER+ Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Puma Biotechnology, Inc. (Industry)
Responsible Party: Principal Investigator, Jose Pablo Leone, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-318
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neratinib (Experimental): * Neratinib will be administered orally once daily
  * Neratinib is dosed at 240mg (six 40mg tablets)
  Interventions: Drug: Neratinib
- Neratinib + Fulvestrant (Experimental): * Neratinib will be administered orally once daily
  * Neratinib is dosed at 240mg (six 40mg tablets)
  * Fulvestrant will be administered intramuscular as an injection (shot) on day 1 and 15 of cycle 1, day 1 of cycle 2, and then on day 1 of each subsequent cycle.
  * Fulvestrant is dosed as 250 mg/5mL (x2) for a total of 500 mg via intramuscular injection (two injections).
  Interventions: Drug: Neratinib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Neratinib — Neratinib is a recently discovered oral drug that may stop breast cancer cells from growing abnormally by inhibiting (or blocking) members of a family of proteins that include Human Epidermal Growth Factor Receptor 2 (HER2)
  Other Names: Nerlynx
Drug: Fulvestrant — Fulvestrant, works in treating breast cancer that has spread to other parts of the body
  Other Names: Faslodex
  Arms: Neratinib + Fulvestrant

SUMMARY:
This research study is studying a drug called Neratinib with and without Fulvestrant as possible treatments for HER2-positive breast cancer .

The interventions involved in this study are:

* Neratinib and Fulvestrant
* Neratinib alone

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has approved Neratinib as a treatment for breast cancer. Fulvestrant has been FDA approved for treatment of metastatic hormone receptor positive breast cancer.

The purpose of this research study is to determine how well neratinib, by itself or together with Fulvestrant, works in treating breast cancer that has spread to other parts of the body. Neratinib is a recently discovered oral drug that may stop breast cancer cells from growing abnormally by inhibiting (or blocking) members of a family of proteins that include Human Epidermal Growth Factor Receptor 2 (HER2).

Neratinib has been used in other research studies and information from those other research studies suggests that neratinib may help to shrink or stabilize HER2-positive breast cancer in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed inoperable locally advanced or metastatic ER+ breast cancer. To fulfill the requirement for ER+ disease, a breast cancer must express, by immunohistochemistry (IHC), ER in ≥10% of cells, on the most recent biopsy. If ER quantification is not available, a determination of ER+ by IHC will suffice. Central confirmation of ER status is not required.
* Participants must have documented HER2+ disease by overexpression and/or gene amplification on the most recent biopsy, per current ASCO-CAP (American Society of Clinical Oncology - College of American Pathologists) guidelines. Central confirmation of HER2 status is not required.
* Participants must have received prior therapy with the following agents in any combination, and in setting (i.e., neoadjuvant, adjuvant, metastatic, etc.). These therapies do not need to be the most recent line of therapy.

  * Trastuzumab
  * Pertuzumab
  * Ado-trastuzumab emtansine (T-DM1)
* Participants must agree to undergo a research biopsy of a reasonably accessible metastatic lesion (chest wall, skin, subcutaneous tissue, lymph nodes, skin, breast, bones, lung, and liver metastases). If a reasonably accessible metastatic lesion is not available, the patient may go on study provided that archived tissue is available. However, if a reasonably accessible site is available for biopsy, the patient must agree to biopsy. Any patients not undergoing biopsy must be approved for study enrollment by the Overall Principal Investigator at DFCI. Biopsies may be done with local anesthesia or intravenous conscious sedation, according to institutional guidelines. If a biopsy requires general anesthesia, then it is only allowed if acquisition of tissue is clinically indicated, and excess tissue may be collected for research purposes. Patients without sites available for biopsy must have available tissue [archived formalin-fixed paraffin embedded blocks (FFPB), blocks from which slides can be created, or fresh frozen tissue from original diagnosis or metastatic setting] for correlative studies. Tissue needs to be located and available at the time of registration See Section 9.3 for more details.
* Women ≥ 18 years of age. Men are not eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (see Appendix A).
* Participants must have normal organ and marrow function as described below:

  * Absolute neutrophil count ≥1,000/uL
  * Platelets ≥75,000/uL
  * Hemoglobin ≥8g/dL
  * Total bilirubin ≤ 1.5 X institutional upper limit of normal (ULN); in case of known Gilbert's syndrome, <2 x ULN is allowed
  * AST(SGOT)/ALT(SGPT) ≤3X institutional ULN without liver metastases, or ≤5X institutional ULN with liver metastases
  * Creatinine clearance ≥ 50 mL/min
  * Left ventricular ejection fraction ≥50%, as determined by RVG (MUGA) or echocardiogram (ECHO) within 60 days prior to initiation of protocol therapy
* Participants may have received any number of prior therapies as long as they have adequate performance status and meet all other eligibility criteria.
* Women of childbearing potential (including premenopausal women and women less than 12 months after menopause) must have a negative β-human chorionic gonadotropin (hCG) urine pregnancy test within 4 weeks of registration.
* The effects of neratinib and fulvestrant on the developing human fetus are unknown. For this reason and because SERD agents are known to be teratogenic, women of child-bearing potential must agree to be abstinent, or to use a highly effective double barrier method of contraception (e.g, a combination of male condom with an intravaginal device such as the cervical cap, diaphragm, or vaginal sponge with spermicide) or a non-hormonal method, while enrolled in the study, until at least 28 days after the last dose of neratinib or 1 year after the last dose of fulvestrant. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately. If a woman is of childbearing potential, she must agree to use adequate contraception prior to the study, for the duration of study participation, and for one year after completion of the study drug.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to neratinib or fulvestrant.
* Participants who have known hypersensitivity to any component of loperamide or colestipol.
* Participants who have received previous therapy with neratinib.
* Participants who have received anti-cancer therapy (including chemotherapy, biological therapy, investigational agents, hormonal therapy, or other anti-cancer therapy) or radiotherapy within ≤14 days prior to the planned initiation of investigational products, or those who have not recovered to grade ≤1from adverse events due to their most recent therapy (excepting alopecia).
* Participants who have had any major surgery ≤28 days prior to the planned initiation of study therapy, or those who have not recovered from adverse events due to agents/surgery administered more than 4 weeks earlier.
* Participants who are receiving any other investigational agents.
* Participants with known brain metastases that are untreated, symptomatic, or require therapy to control symptoms. Participants with a history of treated central nervous system (CNS) metastases are eligible. Treated brain metastases are defined as those without ongoing requirement for corticosteroids, as ascertained by clinical examination and/or brain imaging (magnetic resonance imaging or CT scan) completed during screening. Any corticosteroid use for brain metastases must have been discontinued without the subsequent appearance of symptoms for ≥ 7 days prior to registration. Treatment for brain metastases may include whole brain radiotherapy, radiosurgery, surgery or a combination as deemed appropriate by the treating physician. Radiation therapy must be completed at least 14 days prior to registration.
* Participant has active, uncontrolled cardiac disease, including cardiomyopathy, congestive heart failure (New York Heart Association functional classification of ≥2), unstable angina, myocardial infarction within 12 months of enrollment, or ventricular arrhythmia.
* Participant has a QTc interval >470 ms or known history of QTc prolongation or Torsade de Pointes.
* Participant has an active infection or unexplained fever >38.5°C (101.3°F).
* Participant has had another malignancy within the past 5 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the breast, cervix or vulva; or c) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder, or benign tumors of the adrenal or pancreas.
* Participant has significant chronic gastrointestinal disorder with diarrhea as a major symptom (e.g., Crohn's disease, malabsorption, or Grade ≥2 (NCI CTCAE v.4.0) diarrhea of any etiology at screening).
* Participant has known active infection with hepatitis B or hepatitis C virus. Hepatitis B and C serology testing is not required, unless active infection is suspected.
* Participant is unable or unwilling to swallow tablets.
* Participant has evidence of significant medical illness, abnormal laboratory finding, or psychiatric illness/social situations that would, in the Investigator's judgment, limit compliance with study requirements.
* Pregnant women are excluded from this study because fulvestrant is a SERD agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with neratinib and/or fulvestrant, breastfeeding should be discontinued if the mother is treated with neratinib and/or fulvestrant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Leone, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Indiana University, Indianapolis, Indiana
  - Eastern Maine Medical Center, Brewer, Maine
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber/New Hampshire Oncology-Hematology, Londonderry, New Hampshire
  - The Ohio State University, Columbus, Ohio
  - UT Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Neratinib: * Neratinib will be administered orally once daily
  * Neratinib is dosed at 240mg (six 40mg tablets)
  Neratinib: Neratinib is a recently discovered oral drug that may stop breast cancer cells from growing abnormally by inhibiting (or blocking) members of a family of proteins that include Human Epidermal Growth Factor Receptor 2 (HER2)
- Neratinib + Fulvestrant: * Neratinib will be administered orally once daily
  * Neratinib is dosed at 240mg (six 40mg tablets)
  * Fulvestrant will be administered intramuscular as an injection (shot) on day 1 and 15 of cycle 1, day 1 of cycle 2, and then on day 1 of each subsequent cycle.
  * Fulvestrant is dosed as 250 mg/5mL (x2) for a total of 500 mg via intramuscular injection (two injections).
  Neratinib: Neratinib is a recently discovered oral drug that may stop breast cancer cells from growing abnormally by inhibiting (or blocking) members of a family of proteins that include Human Epidermal Growth Factor Receptor 2 (HER2)
  Fulvestrant: Fulvestrant, works in treating breast cancer that has spread to other parts of the body
Period: Overall Study
Arm/Group | Neratinib | Neratinib + Fulvestrant
Started | 11 | 10
Completed | 10 | 8
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Became ineligible prior to treatment start | 0 | 1
Not completed — progressed before treatment start | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population is only including treated patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Neratinib | Neratinib + Fulvestrant | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Median (Full Range); unit: years] | 55 [28 to 73] | 55.5 [36 to 66] | 55 [28 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 8 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 0 | 2 | 2
  Race: Black or African American | 1 | 0 | 1
  Race: Other | 1 | 0 | 1
  Race: White | 8 | 6 | 14
Prior use of Fulvestrant [Count of Participants; unit: Participants]
  Yes | 3 | 0 | 3
  No | 7 | 8 | 15
Prior lines of therapy [Count of Participants; unit: Participants]
  Less than or equal to 3 lines | 1 | 1 | 2
  Greater than 3 lines | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression-Free Survival (PFS) is defined as the time from randomization (or registration) to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Disease assessment were conducted at baseline and every two cycles after the first cycle.
Time Frame: Participants were followed for PFS up to 20.3 months from registration.
Population: Only treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neratinib | Neratinib + Fulvestrant
Number analyzed (Participants) | 10 | 8
months
  Less than 4 prior lines of therapy; no prior use of fulvestrant: number analyzed (Participants) | 1 | 1
  Less than 4 prior lines of therapy; no prior use of fulvestrant | 19.58 [NA to NA] — The sample size for this group is too small to have a valid interval. | 1.74 [NA to NA] — The sample size for this group is too small to have a valid interval.
  More than 3 prior lines of therapy; no prior use of fulvestrant: number analyzed (Participants) | 7 | 7
  More than 3 prior lines of therapy; no prior use of fulvestrant | 1.81 [1.81 to NA] — The sample size for this group is too small to have a valid interval. | 3.84 [1.61 to NA] — The sample size for this group is too small to have a valid interval.
  More than 3 prior lines of therapy; prior use of fulvestrant: number analyzed (Participants) | 2 | 0
  More than 3 prior lines of therapy; prior use of fulvestrant | 6.42 [5.55 to NA] — The sample size for this group is too small to have a valid interval. |
Statistical Analysis 1: Comparison: Neratinib vs Neratinib + Fulvestrant; Test type: Superiority; p = 0.98, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.27 to 4.12]

2. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive. Participants will be evaluated every 6 months for survival until death. Participants removed from protocol therapy for unacceptable adverse event(s) will be followed until resolution or stabilization of the adverse event.
Time Frame: Participants were followed for up to 38.4 months (3 years and 2 months) from registration to removal from protocol therapy or death.
Population: Only included the treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neratinib | Neratinib + Fulvestrant
Number analyzed (Participants) | 10 | 8
months
  Less than 4 prior lines of therapy; no prior fulvestrant use: number analyzed (Participants) | 1 | 1
  Less than 4 prior lines of therapy; no prior fulvestrant use | NA [NA to NA] — Did not reach median survival. | 12.22 [NA to NA] — Sample size too small to get a valid confidence interval.
  More than 3 prior lines of therapy; no prior fulvestrant use: number analyzed (Participants) | 7 | 7
  More than 3 prior lines of therapy; no prior fulvestrant use | 20.17 [12.91 to NA] — Sample size too small to get a valid confidence interval. | 19.91 [13.63 to NA] — Sample size too small to get a valid confidence interval.
  More than 3 prior lines of therapy; prior fulvestrant use: number analyzed (Participants) | 2 | 0
  More than 3 prior lines of therapy; prior fulvestrant use | 27.79 [NA to NA] — Sample size too small to get a valid confidence interval. |
Statistical Analysis 1: Comparison: Neratinib vs Neratinib + Fulvestrant; Test type: Superiority; p = 0.89, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.24 to 2.81]

3. Secondary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR; Overall Response Rate(ORR) = (CR + PR)/sample size.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib | Neratinib + Fulvestrant
Number analyzed (Participants) | 10 | 8
Participants | 0 | 1

4. Secondary Outcome: Duration Of Responses
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause. Participants without events reported are censored at the last disease evaluation).
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Neratinib | Neratinib + Fulvestrant
Number analyzed (Participants) | 10 | 8
months | NA [NA to NA] — No patient had a response. | 6.7 [NA to NA] — There was only one patient who had a response. The duration of response is 6.7 months.

ADVERSE EVENTS:
Time Frame: 38.4 months (3 years and 2 months)
Arm/Group | Neratinib | Neratinib + Fulvestrant
All-Cause Mortality (participants affected / at risk) | 6/10 | 7/8
Serious Adverse Events (participants affected / at risk) | 4/10 | 2/8
Other Adverse Events (participants affected / at risk) | 10/10 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib (N=10) | Neratinib + Fulvestrant (N=8)
Diarrhea (Gastrointestinal disorders) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Fatigue (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
CPK increased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Bladder perforation (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib (N=10) | Neratinib + Fulvestrant (N=8)
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 7 | 5
Diarrhea (Gastrointestinal disorders) | 8 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 4
Oral pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 6 | 5
Fever (General disorders) | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1
Pain (General disorders) | 4 | 4
Portal hypertension (Hepatobiliary disorders) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2
Alkaline phosphatase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 2
Lymphocyte count decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 2 | 2
Insomnia (Psychiatric disorders) | 2 | 2
Dyspareunia (Reproductive system and breast disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 | 1
Hot flashes (Vascular disorders) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Bronchial infection (Infections and infestations) | 1 | 0
Papulopustular rash (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Investigations - Other, specify (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Hematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT03289039/Prot_SAP_000.pdf